CLINICAL TRIAL: NCT01842633
Title: A Study to Assess Efficacy Over Placebo and Speed of Onset of Pain Relief of New Paracetamol and Caffeine Tablets as Compared to Ibuprofen in Episodic Tension Type Headache
Brief Title: Clinical Study to Evaluate Efficacy of New Paracetamol Formulation Compared to Ibuprofen in Headache
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202172; RH01649 (Other: GSK)
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Caffeine; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paracetamol/ Caffeine Caplets (Experimental): Two caplets of paracetamol/caffeine combination plus 2 placebo caplets to be administered
  Interventions: Drug: Paracetamol and Caffeine
- Ibuprofen Caplets (Active Comparator): Two ibuprofen caplets plus two placebo caplets to be administered
  Interventions: Drug: Ibuprofen
- Placebo Caplets (Placebo Comparator): Four placebo caplets to be administered
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Paracetamol and Caffeine — Caplets containing 500 milligrams (mg) of paracetamol and 65 mg of caffeine
  Arms: Paracetamol/ Caffeine Caplets
Drug: Ibuprofen — Caplets containing 200 mg of ibuprofen
  Arms: Ibuprofen Caplets
Other: Placebo — Matching placebo caplets
  Arms: Placebo Caplets

SUMMARY:
The purpose of this multi-center study is to assess the efficacy of headache relief of new paracetamol/caffeine formulation compared to placebo and ibuprofen in episodic tension-type headache (ETTH).

ELIGIBILITY:
Inclusion Criteria:

* Participants in good general health, and with diagnosis of ETTH with following conditions:

  1. number of days with the condition is historically greater than or equal to two per month;
  2. severity of headaches is historically at least moderate;
  3. duration of headaches is historically more than or equal to 4 hours, if untreated.

     Exclusion Criteria:
* Participant with known or suspected hypersensitivity, allergy, intolerance or contraindication to the use of any of the study medications
* Participant has chronic tension type headache, psychiatric disease or a significant cognitive disorder, or any chronic pain disorder.
* Participant currently taking or has taken medications or herbal supplements within the three months that are likely to interfere with the validity of subject-rated assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- PAREXEL International, LLC, Waltham, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at clinical sites in the United States.
Pre-assignment Details: 365 participants were enrolled in the study out of which 165 participants were randomized in the study. 200 participants were not randomized for the following reasons: 165 were screening failure, 3 due to Adverse Events (AEs), 7 were lost to follow-up, 19 withdrawals by participant, and 6 due to other reasons.
Groups:
- Paracetamol/ Caffeine Caplets: Participants were administered with two caplets of paracetamol/caffeine combination 500/65milligram (mg) plus 2 placebo caplets orally with 8 ounces of water
- Ibuprofen Caplets: Participants were administered with two caplets of ibuprofen 200mg plus 2 placebo caplets orally with 8 ounces of water
- Placebo Caplets: Participants were administered with four placebo caplets with 8 ounces of water
Period: Overall Study
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Started | 65 | 66 | 34
Completed | 62 | 64 | 34
Not Completed | 3 | 2 | 0
Not completed — Screen Failure | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Technical issues | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demography data is available for 157 Participants only (safety Population).
Groups:
- Paracetamol/ Caffeine Caplets: Participants were administered with two caplets of paracetamol/caffeine combination 500/65mg plus 2 placebo caplets orally with 8 ounces of water
- Placebo Caplets: Participants were administered with four placebo caplets orally with 8 ounces of water
- Total: Total of all reporting groups
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets | Total
Number analyzed (Participants) | 62 | 62 | 33 | 157
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.9 (11.39) | 38.1 (13.13) | 38.5 (12.65) | 38.9 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 44 | 23 | 113
  Male | 16 | 18 | 10 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 4 | 14
  White | 56 | 55 | 28 | 139
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID) of Treatment and Placebo at 4 Hours
Description: SPID was calculated as the weighted sum of Pain (Headache) intensity differences at 4 hours post dose. The time-intervals used were 0-10, 10-15, 15-20, 20-25, 25-30, 30-40, 40-50, 50-60, 60-90, 90-120, 120-180, 180-240 minutes. The range of SPID at 4 hours post dose was from -12 to 4". PID was calculated as difference of pain intensity (PI) at baseline (prior to the first dose) with PI at a given time point. PI was assessed on a 4-point scale (0-no headache, 1-mild headache, 2-moderate headache, 3-severe headache).
Time Frame: Up to 4 hours post dose
Population: Intention-to-treat (ITT) population defined as all participants who received treatment and who had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Paracetamol/ Caffeine Caplets: Participants were administered with two caplets of paracetamol/caffeine combination 500/65mg plus two placebo caplets orally with eight ounce of water
- Ibuprofen Caplets: Participants were administered with two caplets of ibuprofen 200mg plus two placebo caplets orally with eight ounce of water
- Placebo Caplets: Participants were administered with four placebo caplets orally with eight ounce of water
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
score on a scale | -6.13 (2.164) | -5.78 (2.098) | -5.86 (2.339)
Statistical Analysis 1: Comparison: Paracetamol/ Caffeine Caplets vs Placebo Caplets; Test type: Superiority or Other; Treatment Difference = -0.47, 95% CI 2-sided [-1.36 to 0.42]

2. Secondary Outcome: Sum of Pain Intensity Difference (SPID) at 1, 2 and 3 Hours
Description: SPID was calculated as the weighted sum of Pain (Headache) intensity differences at 1, 2 and 3 hours post dose.
  The time-intervals used were 0-10, 10-15, 15-20, 20-25, 25-30, 30-40, 40-50, 50-60 minutes for SPID at 1 hour post dose. The range of SPID at 1 hour post dose was from -3 to 1. The time-intervals used were 0-10, 10-15, 15-20, 20-25, 25-30, 30-40, 40-50, 50-60, 60-90, 90-120 minutes for SPID at 2 hours post dose . The range of SPID at 2 hours post dose was from -6 to 2. The time-intervals used were 0-10, 10-15, 15-20, 20-25, 25-30, 30-40, 40-50, 50-60, 60-90, 90-120, 120-180 minutes for SPID at 3 hours post dose. The range of SPID at 3 hours post dose was from -9 to 3. PID was calculated as difference of pain intensity (PI) at baseline (prior to the first dose) with PI at a given time point. PI was assessed on a 4-point scale (0-no headache, 1-mild headache, 2-moderate headache, 3-severe headache).
Time Frame: From (Baseline) 0 to 1 hour, 0 to 2 hours, and 0 to 3 hours post dose
Population: ITT population defined as all participants who received treatment and who had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
score on a scale
  At 1 hour (n=62, 61, 33) | -0.64 (0.488) | -0.56 (0.418) | -0.57 (0.505)
  At 2 hour (n=62, 61, 33) | -2.21 (1.106) | -2.02 (1.002) | -2.04 (1.088)
  At 3 hour (n=61, 62, 32) | -4.09 (1.524) | -3.86 (1.342) | -3.97 (1.528)

3. Secondary Outcome: Number of Participants With Perceptible Pain Relief
Time Frame: Baseline up to 4 hours
Population: as for outcome 2
Measure: Number; unit: number of participants
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
number of participants
  number of participants | 62 | 61 | 33
  number of censored participants | 0 | 1 | 0

4. Secondary Outcome: Time to Perceptible Headache Relief
Description: Time to perceptible headache relief was assessed as the time when participants achieve pain relief scores (PRS) more than or equal to 1.
Time Frame: Baseline up to 4 hours
Population: as for outcome 2
Measure: Median (Full Range); unit: minutes (min.)
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
minutes (min.) | 27.00 (31.274) [6.0 to 140.3] | 29.67 (41.173) [8.7 to 240.0] | 27.00 (38.042) [4.0 to 156.7]

5. Secondary Outcome: Number of Participants With Meaningful Pain Relief
Time Frame: Baseline up to 4 hours
Population: as for outcome 2
Measure: Number; unit: number of participants
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
number of participants
  number of participants | 61 | 60 | 32
  number of censored participants | 1 | 2 | 1

6. Secondary Outcome: Time to Meaningful Headache Relief
Description: Time to meaningful headache relief was assessed as time when participants reported a PRS ≥ 2.
Time Frame: Baseline up to 4 hours
Population: as for outcome 2
Measure: Median (Full Range); unit: min.
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
min. | 43.33 (49.342) [11.7 to 240.0] | 54.17 (49.095) [16.7 to 240.0] | 46.67 (61.477) [12.5 to 240.0]

7. Secondary Outcome: Total Pain Relief (TOTPAR)
Description: TOTPAR was calculated as the weighted sum of pain relief scores (PRS) at each time point. PRS was assessed on a 5-point scale (0-no relief, 1-a little relief, 2-some relief, 3-a lot of relief, and 4-complete relief). The range for TOTPAR for different time points were as follows: from 0 to 4 for TOTPAR at 1 hour post dose, from 0 to 8 for TOTPAR at 2 hours post dose, from 0 to 12 for TOTPAR at 3 hours post dose, and from 0 to 16 for TOTPAR at 4 hours post dose.
Time Frame: From (Baseline) 0 to 1, from 0 to 2, from 0 to 3 and from 0 to 4 hour post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
score on a scale
  Baseline-1 hour (62, 61, 33) | 1.31 (0.922) | 1.17 (0.801) | 1.14 (0.864)
  Baseline-2 hour (62, 61, 33) | 4.28 (1.818) | 4.05 (1.740) | 3.82 (1.886)
  Baseline-3 hour (61, 62, 33) | 7.84 (2.337) | 7.51 (2.250) | 7.35 (2.463)
  Baseline-4 hour (59, 59, 33) | 11.57 (3.373) | 11.05 (3.774) | 10.47 (4.053)

8. Secondary Outcome: Area Under the Time-Response Curve for Change in Headache Intensity and Headache Relief (SPRID)
Description: SPRID was measured as sum of TOTPAR and SPID. SPID and TOTPAR were calculated as weighted sums of PID and PRS at each measurement time point, respectively. PID at each time point was calculated as difference of PI at baseline (prior to the first dose) with PI at a given time point. PI was assessed on a 4-point scale (0-no headache, 1-mild headache, 2-moderate headache, 3-severe headache). PRS was assessed on a 5-point scale (0-no relief, 1-a little relief, 2-some relief, 3-a lot of relief, and 4-complete relief). The range of SPRID for different time points were as follow: from-3 to 5 for SPRID at 1 hour post dose, from -6 to 10 for SPRID at 2 hours post dose, from -9 to 15 for SPRID at 3 hours post dose, and from -12 to 20 for SPRID at 4 hours post dose.
Time Frame: From (Baseline) 0 to 1 hour, 0 to 2 hours, 0 to 3 hours and 0 to 4 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
score on a scale
  At 1 hour (n=62, 61, 33) | 0.67 (0.505) | 0.61 (0.424) | 0.57 (0.473)
  At 2 hour (n=62, 61, 33) | 2.07 (0.957) | 2.03 (0.933) | 1.78 (1.116)
  At 3 hour (n=61, 62, 32) | 3.75 (1.250) | 3.64 (1.285) | 3.38 (1.581)
  At 4 hour (n=59, 59, 33) | 5.44 (1.890) | 5.28 (2.126) | 4.61 (2.613)

9. Secondary Outcome: Global Evaluation of Response to Treatment
Description: Global evaluation of treatment response was measured by a score in a scale from: 0-very poor, 1-poor, 2-neutral [neither poor nor good], 3-good, or 4-very good).
Time Frame: 4 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
score on a scale | 2.88 (0.740) | 2.81 (0.834) | 2.66 (0.946)

10. Secondary Outcome: Rate of Rescue Medication
Description: Number of participants that took rescue medication over the total number of participants for a given treatment group
Time Frame: 4 hours
Population: ITT population defined as all participants who received treatment, who took rescue medication and who had at least one post-baseline efficacy assessment.
Measure: Number; unit: number of participants
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
number of participants | 2 | 4 | 4

11. Secondary Outcome: Change From Baseline in Headache Pain Intensity
Description: Change from baseline in headache pain intensity was calculated as the change (difference) from baseline PI with PI at each time-point. PI was assessed on a 4-point scale (0-no headache, 1-mild headache, 2-moderate headache, 3-severe headache).
Time Frame: At 10, 15, 20, 25, 30, 40, 50, 60, 90, 120, 180, and 240 min.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
score on a scale
  At 10 min. | -0.03 (0.166) | -0.01 (0.064) | -0.04 (0.211)
  At 15 min. | -0.10 (0.322) | -0.06 (0.208) | -0.10 (0.366)
  At 20 min. | -0.27 (0.439) | -0.21 (0.359) | -0.21 (0.464)
  At 25 min. | -0.45 (0.501) | -0.34 (0.438) | -0.36 (0.582)
  At 30 min. | -0.66 (0.625) | -0.51 (0.531) | -0.55 (0.697)
  At 40 min. | -0.92 (0.727) | -0.75 (0.618) | -0.75 (0.729)
  At 50 min. | -1.07 (0.769) | -0.93 (0.736) | -0.96 (0.725)
  At 60 min. | -1.26 (0.831) | -1.17 (0.751) | -1.14 (0.706)
  At 90 min. | -1.51 (0.748) | -1.48 (0.708) | -1.39 (0.733)
  At 120 min. | -1.76 (0.704) | -1.73 (0.727) | -1.69 (0.725)
  At 180 min. | -1.95 (0.529) | -1.90 (0.530) | -1.93 (0.561)
  At 240 min. | -2.01 (0.575) | -1.91 (0.609) | -1.95 (0.591)

12. Secondary Outcome: Headache Relief
Description: The participant assessed headache relief of each treated qualifying headache at 10, 15, 20, 25, 30, 40, 50, 60, 90, 120, 180, and 240 minutes post treatment on a 5-point scale (0-no relief, 1-a little relief, 2-some relief, 3-a lot of relief, and 4-complete relief). higher headache relief score indicates better outcome.
Time Frame: At 10 min. 15 min., 20 min., 25 min., 30 min., 40 min., 50 min., 60 min., 90 min., 120 min., 180 min., 240 min.,
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Paracetamol/ Caffiene Caplets: Participants were administered with two caplets of paracetamol/caffeine combination 500/65mg plus two placebo caplets orally with eight ounce of water
Arm/Group | Paracetamol/ Caffiene Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
score on a scale
  10 min. | 0.07 (0.301) | 0.03 (0.140) | 0.11 (0.379)
  15 min. | 0.33 (0.660) | 0.16 (0.374) | 0.27 (0.635)
  20 min. | 0.68 (0.870) | 0.49 (0.670) | 0.60 (0.876)
  25 min. | 1.06 (1.059) | 0.77 (0.870) | 0.88 (0.986)
  30 min. | 1.37 (1.158) | 1.17 (1.072) | 1.22 (1.107)
  40 min. | 1.86 (1.341) | 1.62 (1.195) | 1.49 (1.182)
  50 min. | 2.15 (1.404) | 1.91 (1.356) | 1.82 (1.218)
  60 min. | 2.42 (1.380) | 2.34 (1.255) | 2.14 (1.213)
  90 min. | 2.85 (1.249) | 2.91 (1.162) | 2.68 (1.196)
  120 min. | 3.35 (0.962) | 3.37 (1.113) | 3.03 (1.206)
  180 min. | 3.69 (0.749) | 3.59 (0.907) | 3.44 (0.978)
  240 min. | 3.72 (0.795) | 3.55 (1.138) | 3.32 (1.155)

13. Secondary Outcome: Number of Pain Free Participants
Description: Number of participants with complete relief was calculated as the number of participants who reported PRS = 4-complete relief at 1 hour and 2 hours post dose.
Time Frame: 1 hour and 2 hour post dose
Population: as for outcome 2
Measure: Number; unit: number of participants
Groups:
- Paracetamol/Caffeine Caplets: Participants were administered with two caplets of paracetamol/caffeine combination 500/65mg plus two placebo caplets orally with eight ounce of water
Arm/Group | Paracetamol/Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
number of participants
  At 1 hour | 18 | 17 | 6
  At 2 hour | 38 | 41 | 20

14. Secondary Outcome: Time to the Use of Rescue Medication.
Description: Time taken by the participants to use the rescue medication
Time Frame: Up to 4 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Number analyzed (Participants) | 62 | 62 | 33
Minutes | 239.00 (6.86) | 235.14 (24.06) | 235.55 (12.8)

ADVERSE EVENTS:
Groups:
- Paracetamol/ Caffeine Caplets: Participants were administered with two caplets of paracetamol/caffeine combination 500/65mg plus 2 placebo caplets orally with 8 ounce of water
- Ibuprofen Caplets: Participants were administered with two caplets of ibuprofen 200mg plus 2 placebo caplets orally with 8 ounce of water
- Placebo Caplets: Participants were administered with four placebo caplets orally with 8 ounce of water
Arm/Group | Paracetamol/ Caffeine Caplets | Ibuprofen Caplets | Placebo Caplets
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62 | 0/33
Other Adverse Events (participants affected / at risk) | 4/62 | 3/62 | 1/33
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paracetamol/ Caffeine Caplets (N=62) | Ibuprofen Caplets (N=62) | Placebo Caplets (N=33)
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
HYPOTHYROIDISM (Endocrine disorders) | 1 | 0 | 0
FEELING JITTERY (General disorders) | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PARANASAL SINUS DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Enrollment into the trial was terminated after randomization of 62% of the plan resulting in a significant reduction in study power. The originally planned inferential statistics (p-values) were therefore not presented in tables summarizing results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.